CLINICAL TRIAL: NCT06429436
Title: Vending Machine Naloxone Distribution for Your Community (VENDY): Increasing Reach and Implementation of Naloxone Distribution
Brief Title: Vending Machine Naloxone Distribution for Your Community (VENDY)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Southern Colorado Harm Reduction Association (Unknown); Denver Health and Hospital Authority (Other); Summit County Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0546
Record Dates: First submitted 2024-05-10; First posted 2024-05-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Harm Reduction; Naloxone; Opioid Overdose
MeSH Terms: conditions — Harm Reduction; Opiate Overdose

STUDY DESIGN:
Intervention Model Description: We will be using an interrupted time series design to evaluate naloxone distribution before and after vending machine implementation in each community.
Masking Description: There will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VENDY (Experimental): Each participating site will install at least 1 machine (vending or kiosks) in the respective community for naloxone distribution.
  Interventions: Behavioral: VENDY

INTERVENTIONS:
Behavioral: VENDY — At least 1 machine (vending machine like a snack machine or a machine like a newspaper kiosk) will be placed in the respective community served by the participating organizations. Any person in the community can get naloxone from the machine. The vending machine will require a code that will be placed on the machine for anyone to use. The kiosks are a box that you simply pull open and naloxone can be obtained. Naloxone kits will be provided for free as part of the current naloxone distribution program within each respective organization.

SUMMARY:
Vending machines are an innovative strategy shown to increase access to naloxone, a medication used to reverse opioid overdose. The aim of this proposal is to study the reach of a community-initiated, stakeholder engaged adaptation of naloxone distribution, VEnding machine Naloxone Distribution for Your community (VENDY) program.

DETAILED DESCRIPTION:
This pilot assessment of the VENDY program will take place in 3 communities. Each community will have a machine (vending or kiosks) in which naloxone will be distributed for free to community members. Our preliminary work identified the locations desired by community members who use illegal drugs for machine placement. The pilot test test will include evaluation of the reach (naloxone distribution), adoption (% of sites and staff implementing), and implementation (fidelity to restocking and maintenance protocol) of VENDY in each community.

ELIGIBILITY:
Inclusion Criteria:

* Any person in the community who desires to obtain naloxone will be able to use the machines

Exclusion Criteria:

* Inability to enter a code on a vending machine or open a kiosk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reach | the 6 months pre VENDY implementation and the 6 months post VENDY implementation
  Reach will be assessed using monthly counts of naloxone distribution in the 6 months before and after VENDY implementation. Naloxone counts will include distribution from all sources within the organization and captured through pharmacy fills from the electronic health record and distribution tracking logs. Naloxone machine distribution will be added to the total monthly count in the post implementation phase and obtained using the vending machine electronic software (reporting date and time of distribution) or (for kiosks) the staff monthly refill tracking log capturing quantity of naloxone kits required to fill the machine (captured at least monthly).

SECONDARY OUTCOMES:
Adoption | At the end of program development (program development is the first phase in which each site is developing VENDY over a 6-18 month period of time)
  Adoption is the percentage of sites placing a naloxone vending machine in the respective community that is made available for community members to obtain naloxone.
Fatal Opioid Overdose Events-Effectiveness | pre-implementation in the year prior to a live VENDY program and post implementation in the year following live VENDY program
  The count of fatal opioid overdose events for each respective county in which the participating organization and vending machine reside in the year before and year after VENDY implementation. Overdose will be captured from publicly available data from death records reported by the Colorado Department of Public Health and Environment. To address temporality we will include fatal opioid overdose deaths in a comparison community matching community features (urban/rural status, community population, and opioid death rate).
Fidelity-Implementation | the 6 months following VENDY implementation
  Fidelity is the percentage of time staff refill and maintain the machine per protocol as measured by the vending machine software and machine activity tracking log.
Maintenance | the 6 months following the initial implementation phase (6 months)
  Number of months each organization implementing VENDY continues to make naloxone available in the machines for the 6 months following the initial implementation phase (6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Wagner, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Denver Health, Denver, Colorado
  - Summit County Public Health Department, Frisco, Colorado
  - Southern Colorado Harm Reduction Association, Pueblo, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.